CLINICAL TRIAL: NCT03985943
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Nemolizumab in Subjects With Moderate-to-Severe Atopic Dermatitis
Brief Title: Efficacy and Safety of Nemolizumab in Subjects With Moderate-to-Severe Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.06.SPR.118161
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Moderate-to-Severe Atopic Dermatitis
Keywords: CD14152; Nemolizumab; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — nemolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Nemolizumab (Experimental): Nemolizumab Active
  Interventions: Drug: Nemolizumab

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Nemolizumab — Nemolizumab
  Other Names: CD14152
  Arms: Nemolizumab

SUMMARY:
The main purpose of the study was to assess the efficacy and safety of nemolizumab after a 16-week treatment period in adult and adolescent subjects with moderate-to-severe atopic dermatitis (AD) not adequately controlled with topical treatments.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled, multi-center, parallel-group study in adult and adolescent subjects of age 12 years and above with moderate-to-severe AD. Eligible subjects had a documented history of inadequate response to topical AD medication(s). Approximately 750 subjects were randomized in 2:1 to receive either nemolizumab or placebo, stratified by baseline disease severity (Investigator's Global Assessment (IGA) = 3, moderate; IGA = 4, severe) and peak pruritus numeric rating scale (PP NRS) severity (PP NRS >= 7; PP NRS < 7). A minimum of 250 subjects were randomized in each PP NRS strata. All nemolizumab-treated subjects who were clinical responders at Week 16 (i.e., the end of initial treatment [Initial Treatment Period]/beginning of Maintenance Period) were re-randomized (1:1:1) to different treatment regimens (nemolizumab injections Q4W or every 8 weeks (Q8W) [with placebo injections at Weeks 20, 28, 36, and 44 to maintain the blind] or placebo Q4W). A clinical responder was defined as a subject at Week 16 with an IGA of 0 (clear) or 1 (almost clear) or a >= 75% improvement in EASI from baseline (EASI-75). All placebo-treated subjects who responded to placebo during the Initial Treatment Period continued to receive placebo Q4W in the Maintenance Period.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects aged greater than and equal to (>=) 12 years at the screening visit.
* Chronic atopic dermatitis (according to American Academy of Dermatology Consensus Criteria) that has been present for at least 2 years before the screening visit.
* Eczema Area and Severity Index (EASI) score >=16 at the screening and baseline visits.
* Investigator Global Assessment (IGA) score >= 3 (scale of 0 to 4) at the screening and baseline visits.
* AD involvement >= 10 percent (%) of body surface area (BSA) at screening and baseline visits.
* Peak Pruritus Numerical Rating Scale (PPNRS) score of at least 4.0 at the screening and baseline visit.
* Documented recent history of inadequate response to topical medications (topical corticosteroids [TCS] with or without Topical calcineurin inhibitors [TCI]).
* Female subjects of childbearing potential (that is, fertile, following menarche and until becoming postmenopausal unless permanently sterile) must agree either to be strictly abstinent throughout the study and for 12 weeks after the last study drug injection, or to use an adequate and approved method of contraception throughout the study and for 12 weeks after the last study drug injection.

Key Exclusion Criteria:

* Body weight (<) 30 kilograms (kg).
* Exacerbation of asthma requiring hospitalization in the preceding 12 months. Uncontrolled asthma in the preceding 3 months.
* Cutaneous infection within 1 week before the baseline visit, any infection requiring treatment with oral or parenteral antibiotics, antivirals, antiparasitics or antifungals within 2 weeks before the baseline visit, or any confirmed or suspected coronavirus disease (COVID)-19 infection within 2 weeks before the screening or baseline visit.
* Pregnant women, breastfeeding women, or women planning a pregnancy during the clinical study.

Note: Subjects with chronic, stable use of prophylactic treatment for recurrent herpes viral infection can be included in this clinical study.

* History of hypersensitivity (including anaphylaxis) to an immunoglobulin product (plasma-derived or recombinant, example, monoclonal antibody) or to any of the study drug excipients.
* Any clinically significant issue, based on investigator judgement.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 941 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2022-08-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (174):
- United States (57):
  - Galderma Investigational Site 8880, North Little Rock, Arkansas
  - Galderma Investigational Site 8578, Cerritos, California
  - Galderma Investigational Site 8636, Fountain Valley, California
  - Galderma Investigational Site 8888, Fullerton, California
  - Galderma Investigational Site 8686, Lomita, California
  - Galderma Investigational Site 8674, Los Angeles, California
  - Galderma Investigational Site 8125, San Francisco, California
  - Galderma Investigational Site 8895, Santa Ana, California
  - Galderma Investigational Site 8608, Santa Monica, California
  - Galderma Investigational Site 8897, Brandon, Florida
  - Galderma Investigational Site 8805, Cape Coral, Florida
  - Galderma Investigational Site 8902, Doral, Florida
  - Galderma Investigational Site 8804, Hialeah, Florida
  - Galderma Investigational Site 8711, Jacksonville, Florida
  - Galderma Investigational Site 8710, Miami, Florida
  - Galderma Investigational Site 8801, Miami, Florida
  - Galderma Investigational Site 8737, Miami, Florida
  - Galderma Investigational Site 8708, Miami, Florida
  - Galderma Investigational Site 8806, Miami Lakes, Florida
  - Galderma Investigational Site 8800, Miami Lakes, Florida
  - Galderma Investigational Site 8734, Pembroke Pines, Florida
  - Galderma Investigational Site 8744, Macon, Georgia
  - Galderma Investigational Site 8728, Newnan, Georgia
  - Galderma Investigational Site 8887, Union City, Georgia
  - Galderma Investigational Site 8890, Blackfoot, Idaho
  - Galderma Investigational Site 8819, Nampa, Idaho
  - Galderma Investigational Site 8571, Skokie, Illinois
  - Galderma Investigational Site 8712, Skokie, Illinois
  - Galderma Investigational Site 8142, Indianapolis, Indiana
  - Galderma Investigational Site 8771, Louisville, Kentucky
  - Galderma Investigational Site 8882, Bangor, Maine
  - Galderma Investigational Site 8743, Ann Arbor, Michigan
  - Galderma Investigational Site 8512, Bay City, Michigan
  - Galderma Investigational Site 8155, Troy, Michigan
  - Galderma Investigational Site 8748, Ypsilanti, Michigan
  - Galderma Investigational Site 8521, Saint Joseph, Missouri
  - Galderma Investigational Site 8718, Missoula, Montana
  - Galderma Investigational Site 8810, Omaha, Nebraska
  - Galderma Investigational Site 8740, Henderson, Nevada
  - Galderma Investigational Site 8242, Brooklyn, New York
  - Galderma Investigational Site 8620, New York, New York
  - Galderma Investigational Site 8279, New York, New York
  - Galderma Investigational Site 8648, Wilmington, North Carolina
  - Galderma Investigational Site 8702, Bexley, Ohio
  - Galderma Investigational Site 8595, Dublin, Ohio
  - Galderma Investigational Site 8206, Norman, Oklahoma
  - Galderma Investigational Site 8857, Oklahoma City, Oklahoma
  - Galderma Investigational Site 8255, Philadelphia, Pennsylvania
  - Galderma Investigational Site 8802, Plymouth Meeting, Pennsylvania
  - Galderma Investigational Site 8736, Charleston, South Carolina
  - Galderma Investigational Site 8818, Rapid City, South Dakota
  - Galderma Investigational Site 8133, Arlington, Texas
  - Galderma Investigational Site 8238, Dallas, Texas
  - Galderma Investigational Site 8827, Dripping Springs, Texas
  - Galderma Investigational Site 8664, Frisco, Texas
  - Galderma Investigational Site 8042, Houston, Texas
  - Galderma Investigational Site 8862, Fairfax, Virginia
- Australia (11):
  - Galderma Investigational Site 5441, Darlinghurst, New South Wales
  - Galderma Investigational Site 5759, Kogarah, New South Wales
  - Galderma Investigational Site 6152, Westmead, New South Wales
  - Galderma Investigational Site 5638, Benowa, Queensland
  - Galderma Investigational Site 6161, Brisbane, Queensland
  - Galderma Investigational Site 6159, Woodville, South Australia
  - Galderma Investigational Site 6131, Carlton, Victoria
  - Galderma Investigational Site 5366, East Melbourne, Victoria
  - Galderma Investigational Site 5458, Parkville, Victoria
  - Galderma Investigational Site 5453, Fremantle, Western Australia
  - Galderma Investigational Site 6153, Victoria Park, Western Australia
- Austria (3):
  - Galderma Investigational Sites 6157, Graz, Styria
  - Galderma Investigational Site 6194, Vienna, Vienna
  - Galderma Investigational Site 6158, Vienna
- Canada (16):
  - Galderma Investigational Site 8085, Calgary, Alberta
  - Galderma Investigational Site 8903, Calgary, Alberta
  - Galderma Investigational Site 8215, Calgary, Alberta
  - Galderma Investigational Site 8088, Edmonton, Alberta
  - Galderma Investigational Site 8824, Edmonton, Alberta
  - Galderma Investigational Site 8722, Edmonton, Alberta
  - Galderma Investigational Site 8161, Surrey, British Columbia
  - Galderma Investigational Site 8586, Barrie, Ontario
  - Galderma Investigational Site 8904, Guelph, Ontario
  - Galderma Investigational Site 8901, Ottawa, Ontario
  - Galderma Investigational Site 8336, Toronto, Ontario
  - Galderma Investigational Site 8899, Toronto, Ontario
  - Galderma Investigational Site 8780, Niagara Falls
  - Galderma Investigational Site 8610, Ottawa
  - Galderma Investigational Site 8000, Saint John
  - Galderma Investigational Site 8731, Waterloo
- Czechia (8):
  - Galderma Investigational Site 6055, Brno
  - Galderma Investigational Site 5225, Náchod
  - Galderma Investigational Site 6030, Olomouc
  - Galderma Investigational Site 6024, Prague
  - Galderma Investigational Site 6054, Prague
  - Galderma Investigational Site 6021, Prague
  - Galderma Investigational Site 6240, Prague
  - Galderma Investigational Site 6025, Prague
- Germany (13):
  - Galderma Investigational Site 6146, Langenau, Hesse
  - Galderma Investigational Site 6214, Tübingen, Niedersachesen
  - Galderma Investigational Site 6172, Berlin, North Rhine-Westphalia
  - Galderma Investigational Site 5437, Kiel, Schleswig-Holst
  - Galderma Investigational Site 6022, Bad Bentheim
  - Galderma Investigational Site 6110, Berlin
  - Galderma Investigational Site 6061, Bielefeld
  - Galderma Investigational Site 6066, Buxtehude
  - Galderma Investigational Site 5368, Darmstadt
  - Galderma Investigational Site 6028, Dülmen
  - Galderma Investigational Site 6039, Münster
  - Galderma Investigational Site 5918, Osnabrück
  - Galderma Investigational Site 6109, Stuttgart
- Latvia (4):
  - Galderma Investigational Site 6113, Liepāja
  - Galderma Investigational Site 6134, Riga
  - Galderma Investigational Site 6059, Riga
  - Galderma Investigational Site 6060, Talsi
- Lithuania (3):
  - Galderma Investigational Site 6111, Kaunas
  - Galderma Investigational Site 6072, Klaipėda
  - Galderma Investigational Site 6112, Vilnius
- Netherlands (3):
  - Galderma Investigational Site 6212, Groningen
  - Galderma Investigational Site 6108, Rotterdam
  - Galderma Investigational Site 6027, Utrecht
- New Zealand (2):
  - Galderma Investigational Site 6119, Hamilton
  - Galderma Investigational Site 6118, Wellington
- Poland (20):
  - Galderma Investigational Site 6255, Częstochowa
  - Galderma Investigational Site 6075, Gdansk
  - Galderma Investigational Site 6243, Gdansk
  - Galderma Investigational Site 5138, Gdansk
  - Galderma Investigational Site 6244, Gdynia
  - Galderma Investigational Site 6087, Katowice
  - Galderma Investigational Site 6245, Lodz
  - Galderma Investigational Site 5570, Lodz
  - Galderma Investigational Site 6231, Lodz
  - Galderma Investigational Site 6071, Lublin
  - Galderma Investigational Site 6237, Ostrowiec Świętokrzyski
  - Galderma Investigational Site 6127, Poznan
  - Galderma Investigational Site 6223, Szczecin
  - Galderma Investigational Site 6065, Warsaw
  - Galderma Investigational Site 6122, Warsaw
  - Galderma Investigational Site 6242, Warsaw
  - Galderma Investigational Site 6064, Warsaw
  - Galderma Investigational Site 6222, Warsaw
  - Galderma Investigational Site 6047, Wroclaw
  - Galderma Investigational Site 5005, Wroclaw
- South Korea (15):
  - Galderma Investigational Site 6095, Bucheon-si
  - Galderma Investigational Site 6100, Busan
  - Galderma Investigational Site 6098, Gyeonggi-do
  - Galderma Investigational Site 6154, Gyeonggi-do
  - Galderma Investigational Site 6138, Incheon
  - Galderma Investigational Site 6120, Incheon
  - Galderma Investigational Site 6093, Incheon
  - Galderma Investigational Site 6105, Seoul
  - Galderma Investigational Site 5659, Seoul
  - Galderma Investigational Site 6116, Seoul
  - Galderma Investigational Site 6129, Seoul
  - Galderma Investigational Site 6103, Seoul
  - Galderma Investigational Site 6056, Seoul
  - Galderma Investigational Site 6094, Seoul
  - Galderma Investigational Site 6099, Seoul
- Spain (11):
  - Galderma Investigational Site 6057, Alicante
  - Galderma Investigational Site 6037, Barcelona
  - Galderma Investigational Site 6035, Barcelona
  - Galderma Investigational Site 5580, Barcelona
  - Galderma Investigational Site 6106, Las Palmas de Gran Canaria
  - Galderma Investigational Site 6058, Madrid
  - Galderma Investigational Site 5842, Madrid
  - Galderma Investigational Site 6190, Madrid
  - Galderma Investigational Site 6036, Madrid
  - Galderma Investigational Site 5551, Madrid
  - Galderma Investigational Site 6191, Pamplona
- United Kingdom (8):
  - Galderma Investigational Site 6202, Barnsley
  - Galderma Investigational Site 6207, Blackpool
  - Galderma Investigational Site 6203, Cannock
  - Galderma Investigational Site 6104, Glasgow
  - Galderma Investigational Site 6204, Liverpool
  - Galderma Investigational Site 6121, London
  - Galderma Investigational Site 6205, Manchester
  - Galderma Investigational Site 6206, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silverberg JI, Filipenko D, Dias Barbosa C, Rodriguez D, Chambenoit O, Jack K, Piketty C, Subramanian R, Puelles J. Patients' Experiences of Atopic Dermatitis and Nemolizumab Treatment: An In-Trial Interview Study Embedded in a Phase 3 Clinical Trial (ARCADIA). Patient. 2025 Sep;18(5):511-521. doi: 10.1007/s40271-025-00741-x. Epub 2025 May 13. PMID 40360966
- [Derived] Silverberg JI, Rodriguez DN, Dias-Barbosa C, Filipenko D, Ulianov L, Piketty C, Puelles J. Psychometric Validation of the Subject Sleep Diary in Patients with Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2025 Apr;15(4):963-995. doi: 10.1007/s13555-025-01385-3. Epub 2025 Mar 21. PMID 40116983
- [Derived] Silverberg JI, Wollenberg A, Reich A, Thaci D, Legat FJ, Papp KA, Stein Gold L, Bouaziz JD, Pink AE, Carrascosa JM, Rewerska B, Szepietowski JC, Krasowska D, Havlickova B, Kalowska M, Magnolo N, Pauser S, Nami N, Sauder MB, Jain V, Padlewska K, Cheong SY, Fleuranceau Morel P, Ulianov L, Piketty C; ARCADIA 1 and ARCADIA 2 Study Investigators. Nemolizumab with concomitant topical therapy in adolescents and adults with moderate-to-severe atopic dermatitis (ARCADIA 1 and ARCADIA 2): results from two replicate, double-blind, randomised controlled phase 3 trials. Lancet. 2024 Aug 3;404(10451):445-460. doi: 10.1016/S0140-6736(24)01203-0. Epub 2024 Jul 24. PMID 39067461
- [Derived] Dias-Barbosa C, Silverberg JI, Stander S, Rodriguez D, Fofana F, Filipenko D, Ulianov L, Piketty C, Puelles J. Capturing patient-reported sleep disturbance in atopic dermatitis clinical trials. J Patient Rep Outcomes. 2024 Jul 15;8(1):73. doi: 10.1186/s41687-024-00751-7. PMID 39008191

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 177 active sites in Australia, Austria, Canada, Czech Republic, Germany, Great Britain, Korea, Latvia, Lithuania, Netherlands, New Zealand, Poland, Spain and the United States from 27 June 2019 to 11 August 2022.
Pre-assignment Details: A total of 941 randomized 2:1 to receive either nemolizumab or placebo.At Week 16, 272 nemolizumab-treated participants were clinical responders (defined as IGA of 0[clear] or 1[almost clear]or Eczema Area and Severity Index [EASI]-75) re-randomized to receive nemolizumab Q4W,nemolizumab Q8W,or placebo during Maintenance Period.100 participants received placebo in Initial Treatment, responded to placebo at Week 16,re-assigned to placebo and continued to receive placebo Q4W in Maintenance Period.
Groups:
- Initial Treatment Period (Baseline - Week 16 Predose): Placebo: Participants received placebo via 2 subcutaneous (SC) injections at Day 1, thereafter, every 4 weeks (Q4W) at Weeks 4, 8, and 12 by a single SC injection during Initial Treatment Period.
- Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg: Participants received nemolizumab 30 milligrams (mg) via 2 SC injections at Day 1, thereafter, Q4W at Weeks 4, 8, and 12 by a single SC injection during Initial Treatment Period.
- Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q4W: Participants who received nemolizumab, Q4W during Initial Treatment Period and were clinical responders (defined as participants with an IGA of 0 (clear) or 1 (almost clear) or a greater than and equal to (>=) 75 percent (%) improvement in EASI from Baseline) at Week 16 received nemolizumab 30 mg, Q4W at Weeks 16, 20, 24, 28, 32, 36, 40, and 44 by a single SC injection during Maintenance Period.
- Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q8W: Participants who received nemolizumab, Q4W during Initial Treatment Period and were clinical responders (defined as participants with an IGA of 0 (clear) or 1 (almost clear) or a >=75% improvement in EASI from Baseline) at Week 16 received nemolizumab 30 mg, every 8 weeks (Q8W) at Weeks 20, 28, 36, and 44 by a single SC injection during Maintenance Period.
- Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Placebo Q4W: Participants who received nemolizumab, Q4W during Initial Treatment Period and were clinical responders (defined as participants with an IGA of 0 (clear) or 1 (almost clear) or a >=75% improvement in EASI from Baseline) at Week 16 received placebo, Q4W at Weeks 16, 20, 24, 28, 32, 36, 40, and 44 by a single SC injection during Maintenance Period.
- Maintenance Period (Week 16-Week 48): Placebo Q4W Re-assigned to Placebo Q4W: Participants who received placebo, Q4W during Initial Treatment Period and were clinical responders (defined as participants with an IGA of 0 (clear) or 1 (almost clear) or a >=75% improvement in EASI from Baseline) at Week 16 received placebo, Q4W at Weeks 16, 20, 24, 28, 32, 36, 40, and 44 by a single SC injection during Maintenance Period.
Period: Initial Treatment(Day 1-Week 16 Predose)
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q4W | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q8W | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Placebo Q4W | Maintenance Period (Week 16-Week 48): Placebo Q4W Re-assigned to Placebo Q4W
Started | 321 | 620 | 0 | 0 | 0 | 0
Safety Population (Safety population (SP) consisted of all participants who received at least 1 dose of study drug.) | 321 | 616 | 0 | 0 | 0 | 0
Completed | 296 | 560 | 0 | 0 | 0 | 0
Not Completed | 25 | 60 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 5 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 9 | 9 | 0 | 0 | 0 | 0
Not completed — Subjects request | 11 | 25 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 10 | 0 | 0 | 0 | 0
Not completed — Protocol deviation | 3 | 4 | 0 | 0 | 0 | 0
Not completed — Physician/Principal Investigators Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Randomized but not treated | 0 | 4 | 0 | 0 | 0 | 0
Period: Maintenance Period (Week 16-Week 48)
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q4W | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q8W | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Placebo Q4W | Maintenance Period (Week 16-Week 48): Placebo Q4W Re-assigned to Placebo Q4W
Started | 0 | 0 | 90 (Participants who received nemolizumab, Q4W during Initial Treatment Period and were clinical responders at Week 16 were re-randomized during Maintenance Period.) | 91 (Participants who received nemolizumab, Q4W during Initial Treatment Period and were clinical responders at Week 16 were re-randomized during Maintenance Period.) | 91 (Participants who received nemolizumab, Q4W during Initial Treatment Period and were clinical responders at Week 16 were re-randomized during Maintenance Period.) | 100 (Participants who received placebo, Q4W during Initial Treatment Period and were clinical responders at Week 16, were re-assigned during Maintenance Period.)
Safety Population | 0 | 0 | 91 (One participant was re-randomized to Nemolizumab Q8W for Maintenance Period, but erroneously received Nemolizumb three times consecutively and thus counted in Nemolizumab 30 mg Q4W to Q4W for safety analysis.) | 90 (One participant was re-randomized to Nemolizumab Q8W for Maintenance Period, but erroneously received Nemolizumb three times consecutively and thus counted in Nemolizumab 30 mg Q4W to Q4W for safety analysis.) | 91 | 100
Completed | 0 | 0 | 76 | 79 | 69 | 82
Not Completed | 0 | 0 | 14 | 12 | 22 | 18
Not completed — Lack of Efficacy | 0 | 0 | 4 | 3 | 12 | 4
Not completed — Adverse Event | 0 | 0 | 1 | 3 | 1 | 1
Not completed — Subjects request | 0 | 0 | 6 | 4 | 5 | 9
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Protocol Deviation | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Physician/PI Decision | 0 | 0 | 2 | 1 | 1 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The ITT population consisted of all randomized participants.
Groups:
- Initial Treatment Period (Baseline - Week 16 Predose): Placebo: Participants received placebo via 2 SC injections at Day 1, thereafter, Q4W at Weeks 4, 8, and 12 by a single SC injection during Initial Treatment Period.
- Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg: Participants received nemolizumab 30 mg via 2 SC injections at Day 1, thereafter, Q4W at Weeks 4, 8, and 12 by a single SC injection during Initial Treatment Period.
- Total: Total of all reporting groups
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Total
Number analyzed (Participants) | 321 | 620 | 941
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (15.61) | 33.5 (15.92) | 33.3 (17.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 297 | 441
  Male | 177 | 323 | 500
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 64 | 96
  Not Hispanic or Latino | 288 | 552 | 840
  Unknown or Not Reported | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 51 | 117 | 168
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 18 | 36 | 54
  White | 244 | 451 | 695
  More than one race | 4 | 10 | 14
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Investigator's Global Assessment (IGA) Success (IGA of 0 or 1 and a More Than Equal to [>=] 2-point Reduction): Intent-To-Treat (ITT) Population
Description: IGA success was defined as an IGA score of 0 (clear) or 1 (almost clear) and at least a 2-grade improvement from baseline to Week 16. The IGA is a 5-point scale ranging from 0 (clear) to 4 (severe) used by the Investigator or trained designee to evaluate the global severity of atopic dermatitis (AD) and the clinical response to treatment. If a participant received any rescue therapy, the data after receipt of rescue therapy was considered treatment failure. Participants with missing data at Week 16 were considered non-responders.
Time Frame: Week 16
Population: The ITT population consisted of all randomized participants. Data was planned to be collected and analyzed for Initial Treatment Period.
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg
Number analyzed (Participants) | 321 | 620
percentage of participants | 24.6 | 35.6
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; A hierarchical testing procedure was used to control the overall type I error. Testing was performed sequentially in order the outcome measures were reported and continued when the test for the preceding outcome measure was statistically significant at two-sided 2.5% significance level; Test type: Other; p = 0.0003, Cochran-Mantel-Haenszel — Strata-adjusted p-values were calculated from Cochran-Mantel-Haenszel test adjusting randomized stratification variables (IGA severity [3=moderate, 4=severe] and PP NRS [>=7, <7]); Strata-adjusted percentage difference = 11.5, 97.5% CI 2-sided [4.7 to 18.3]

2. Primary Outcome: Percentage of Participants With an Investigator's Global Assessment (IGA) Success (IGA of 0 or 1 and a >= 2-point Reduction): Severe Pruritus Population
Description: IGA success was defined as an IGA score of 0 (clear) or 1 (almost clear) and at least a 2-grade improvement from baseline to Week 16. The IGA is a 5-point scale ranging from 0 (clear) to 4 (severe) used by the Investigator or trained designee to evaluate the global severity of AD and the clinical response to treatment. If a participant received any rescue therapy, the data after receipt of rescue therapy was considered a treatment failure. Participants with missing data at Week 16 were considered non-responders.
Time Frame: Week 16
Population: Severe pruritus population consisted of all randomized participants with a baseline PP NRS >=7. Data was planned to be collected and analyzed for Initial Treatment Period.
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg
Number analyzed (Participants) | 210 | 406
percentage of participants | 21.4 | 35.5
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0002, Cochran-Mantel-Haenszel — Strata-adjusted p-values were calculated from Cochran-Mantel-Haenszel test adjusting randomized stratification variables (IGA severity [3=moderate, 4=severe]); Strata-adjusted percentage difference = 14.3, 97.5% CI 2-sided [6.1 to 22.5]

3. Primary Outcome: Percentage of Participants With >=75% Improvement in Eczema Area and Severity Index (EASI-75) at Week 16: ITT Population
Description: EASI-75 was defined as >=75 percent(%) improvement in EASI from baseline to Week 16. EASI evaluates severity of participants AD based on severity of AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD(erythema, induration/papulation, excoriation and lichenification)scored separately for each of 4 body regions (head & neck, upper limbs, trunk & lower limbs on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. If a participant received any rescue therapy, the data after receipt of rescue therapy was considered treatment failure. Participants with missing data at Week 16 were considered non-responders. EASI total score is composite score ranging from 0 to 72. Higher scores represent greater severity of AD.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg
Number analyzed (Participants) | 321 | 620
percentage of participants | 29.0 | 43.5
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 14.9, 97.5% CI 2-sided [7.8 to 22.0]

4. Primary Outcome: Percentage of Participants With >=75% Improvement in Eczema Area and Severity Index (EASI-75) at 16: Severe Pruritus Population
Description: EASI-75 was defined as >=75 percent(%) improvement in EASI from baseline to Week 16. EASI evaluates severity of participants AD based on severity of AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification)scored separately for each of 4 body regions (head & neck, upper limbs, trunk & lower limbs on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. If a participant received any rescue therapy, the data after receipt of rescue therapy was considered treatment failure. Participants with missing data at Week 16 were considered non-responders. EASI total score is composite score ranging from 0 to 72. Higher scores represent greater severity of AD.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg
Number analyzed (Participants) | 210 | 406
percentage of participants | 23.8 | 41.6
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Strata-adjusted percentage difference = 18.1, 97.5% CI 2-sided [9.6 to 26.6]

5. Secondary Outcome: Percentage of Participants With Improvement of >=4 Points in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) at Week 16: ITT Population
Description: The PP NRS is a scale that was used by the participants to report the intensity of their pruritus (itch) during the last 24 hours on a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable'. Weekly average PP NRS score was calculated using 7 consecutive days diary data and set to missing if less than 4 days data available. If a participant received any rescue therapy, the data after receipt of rescue therapy was considered treatment failure.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg
Number analyzed (Participants) | 321 | 620
percentage of participants | 17.8 | 42.7
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; A hierarchical testing procedure was used to control the overall type I error. Testing was performed sequentially in order the outcome measures were reported and continued when the test for the preceding outcome measure was statistically significant at two-sided 2.5% significance level. Participants with missing data were considered non-responders; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 24.9, 97.5% CI 2-sided [18.4 to 31.5]
Statistical Analysis 2: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; Nemolizumab 30 mg versus Placebo using multiple imputation (MI) with missing at random (MAR) assumption; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 28.1, 97.5% CI 2-sided [22.0 to 34.3] — The estimates are from 50 complete datasets by MI-MAR assumption

6. Secondary Outcome: Percentage of Participants With Improvement of >=4 Points in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) at Week 16: Severe Pruritus Population
Description: as for outcome 5
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg
Number analyzed (Participants) | 210 | 406
percentage of participants | 18.6 | 46.1
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; [analysis description as in outcome 5, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — Strata-adjusted p-values were calculated from Cochran-Mantel-Haenszel test adjusting randomized stratification variables (IGA severity [3=moderate, 4=severe]; Strata-adjusted percentage difference = 27.5, 97.5% CI 2-sided [19.4 to 35.7]
Statistical Analysis 2: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; Nemolizumab 30 mg versus Placebo using MI-MAR assumption; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 6, analysis 1]; Strata-adjusted percentage difference = 32.1, 97.5% CI 2-sided [24.4 to 39.8] — The estimates are from 50 complete datasets by MI-MAR assumption

7. Secondary Outcome: Percentage of Participants With <2 Points in Weekly Average PP NRS at Week 16: ITT Population
Description: The PP NRS is a scale that was used by the participants to report the intensity of their pruritus (itch) during the last 24 hours on a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable'. Weekly average PP NRS score was calculated using 7 consecutive days diary data and set to missing if less than 4 days data available. If a participant received any rescue therapy, the data after receipt of rescue therapy was considered treatment failure. Participants with missing data were considered non-responders.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg
Number analyzed (Participants) | 321 | 620
percentage of participants | 11.2 | 30.6
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 19.5, 97.5% CI 2-sided [13.7 to 25.2]

8. Secondary Outcome: Percentage of Participants With <2 Points in Weekly Average PP NRS at Week 16: Severe Pruritus Population
Description: as for outcome 7
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg
Number analyzed (Participants) | 210 | 406
percentage of participants | 7.6 | 27.8
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Strata-adjusted percentage difference = 20.3, 97.5% CI 2-sided [13.8 to 26.8]

9. Secondary Outcome: Percentage of Participants With an Improvement of Sleep Disturbance Numeric Rating Scale (SD NRS) >=4 at Week 16: ITT Population
Description: The sleep disturbance NRS is a scale used by the participants to report the degree of their sleep loss related to AD. Participants were asked the following question in their local language: how would you rate your sleep last night? On a scale of 0 to 10, with 0 being 'no sleep loss related to signs/symptoms of AD' and 10 being 'I cannot sleep at all due to the signs/symptoms of AD'. Weekly average SD NRS score was calculated using 7 consecutive days diary data and set to missing if less than 4 days data available. If a participant received any rescue therapy, the data after receipt of rescue therapy was considered treatment failure. Participants with missing data were considered non-responders.
Time Frame: Week 16
Population: The ITT population consisted of all randomized participants.
Measure: Number; unit: percentage of subjects
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg
Number analyzed (Participants) | 321 | 620
percentage of subjects | 19.9 | 37.9
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 17.9, 97.5% CI 2-sided [11.3 to 24.5]

10. Secondary Outcome: Percentage of Participants With an Improvement of Sleep Disturbance Numeric Rating Scale (SD NRS) >=4 at Week 16: Severe Pruritus Population
Description: as for outcome 9
Time Frame: Week 16
Population: Severe pruritus population consisted of all randomized participants with a baseline PP NRS >=7.
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg
Number analyzed (Participants) | 210 | 406
percentage of participants | 22.4 | 42.1
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Strata-adjusted percentage difference = 19.7, 97.5% CI 2-sided [11.2 to 28.2]

11. Secondary Outcome: Percentage of Participants With Improvement of >=4 Points in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) at Week 4: ITT Population
Description: as for outcome 7
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg
Number analyzed (Participants) | 321 | 620
percentage of participants | 6.5 | 27.4
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 20.9, 97.5% CI 2-sided [15.8 to 26]

12. Secondary Outcome: Percentage of Participants With Improvement of >=4 Points in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) at Week 4: Severe Pruritus Population
Description: as for outcome 7
Time Frame: Week 4
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg
Number analyzed (Participants) | 210 | 406
percentage of participants | 7.1 | 28.3
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Strata-adjusted percentage difference = 21.2, 97.5% CI 2-sided [14.8 to 27.6]

13. Secondary Outcome: Percentage of Participants With Peak Pruritus Numeric Rating Scale (PP NRS) <2 at Week 4: ITT Population
Description: as for outcome 7
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg
Number analyzed (Participants) | 321 | 620
percentage of participants | 3.7 | 16.0
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 12.2, 97.5% CI 2-sided [8.2 to 16.3]

14. Secondary Outcome: Percentage of Participants With Peak Pruritus Numeric Rating Scale (PP NRS) <2 at Week 4: Severe Pruritus Population
Description: as for outcome 7
Time Frame: Week 4
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg
Number analyzed (Participants) | 210 | 406
percentage of participants | 2.9 | 12.6
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Strata-adjusted percentage difference = 9.7, 97.5% CI 2-sided [5.2 to 14.2]

15. Secondary Outcome: Percentage of Participants With Improvement of >=4 Points in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) at Week 2: ITT Population
Description: as for outcome 7
Time Frame: Week 2
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg
Number analyzed (Participants) | 321 | 620
percentage of participants | 3.1 | 17.7
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 14.6, 97.5% CI 2-sided [10.6 to 18.7]

16. Secondary Outcome: Percentage of Participants With Improvement of >=4 Points in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) at Week 2: Severe Pruritus Population
Description: as for outcome 7
Time Frame: Week 2
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg
Number analyzed (Participants) | 210 | 406
percentage of participants | 3.8 | 20.7
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Strata-adjusted percentage difference = 16.9, 97.5% CI 2-sided [11.5 to 22.3]

17. Secondary Outcome: Percentage of Participants With Improvement of >=4 Points in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) at Week 1: ITT Population
Description: as for outcome 7
Time Frame: Week 1
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg
Number analyzed (Participants) | 321 | 620
percentage of participants | 1.2 | 4.5
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0064, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 3.4, 97.5% CI 2-sided [1.1 to 5.8]

18. Secondary Outcome: Percentage of Participants With Improvement of >=4 Points in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) at Week 1: Severe Pruritus Population
Description: as for outcome 7
Time Frame: Week 1
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg
Number analyzed (Participants) | 210 | 406
percentage of participants | 1.9 | 6.2
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Placebo vs Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg; A hierarchical testing procedure was used to control the overall type I error. Testing was performed sequentially in order the outcome measures were reported and continued when the test for preceding outcome measure was statistically significant at two-sided 2.5% significance level; Test type: Other; p = 0.0177, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Strata-adjusted percentage difference = 4.3, 97.5% CI 2-sided [0.9 to 7.7]

ADVERSE EVENTS:
Time Frame: Initial Treatment Period: From baseline to Week 16 pre-dose; Maintenance Period: From end of Initial Treatment Period (i.e., Week 16) to Week 48
Description: The SP comprised all participants who received at least 1 dose of study drug.
Groups:
- Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q4W: Participants who received nemolizumab, Q4W during Initial Treatment Period and were clinical responders (defined as participants with an IGA of 0 (clear) or 1 (almost clear) or a >=75% improvement in EASI from Baseline) at Week 16 received nemolizumab 30 mg, Q4W at Weeks 16, 20, 24, 28, 32, 36, 40, and 44 by a single SC injection during Maintenance Period.
- Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q8W: Participants who received nemolizumab, Q4W during Initial Treatment Period and were clinical responders (defined as participants with an IGA of 0 (clear) or 1 (almost clear) or a >=75% improvement in EASI from Baseline) at Week 16 received nemolizumab 30 mg, every 8 weeks (Q8W) at Weeks 16, 24, 32, and 40 by a single SC injection during Maintenance Period.
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q4W | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q8W | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Placebo Q4W | Maintenance Period (Week 16-Week 48): Placebo Q4W Re-assigned to Placebo Q4W
All-Cause Mortality (participants affected / at risk) | 0/321 | 0/616 | 0/91 | 0/90 | 0/91 | 0/100
Serious Adverse Events (participants affected / at risk) | 4/321 | 6/616 | 4/91 | 3/90 | 2/91 | 1/100
Other Adverse Events (participants affected / at risk) | 67/321 | 144/616 | 27/91 | 28/90 | 33/91 | 35/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Treatment Period (Baseline - Week 16 Predose): Placebo (N=321) | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg (N=616) | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q4W (N=91) | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q8W (N=90) | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Placebo Q4W (N=91) | Maintenance Period (Week 16-Week 48): Placebo Q4W Re-assigned to Placebo Q4W (N=100)
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Splenic injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Periarthiritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Plasmablastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Treatment Period (Baseline - Week 16 Predose): Placebo (N=321) | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg (N=616) | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q4W (N=91) | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q8W (N=90) | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Placebo Q4W (N=91) | Maintenance Period (Week 16-Week 48): Placebo Q4W Re-assigned to Placebo Q4W (N=100)
COVID-19 (Infections and infestations) | 6 | 10 | 9 | 9 | 6 | 10
Nasopharyngitis (Infections and infestations) | 8 | 9 | 7 | 5 | 7 | 6
Upper respiratory tract infection (Infections and infestations) | 14 | 9 | 3 | 3 | 5 | 9
Headache (Nervous system disorders) | 11 | 28 | 5 | 5 | 3 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 13 | 33 | 3 | 6 | 5 | 5
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 33 | 73 | 7 | 8 | 12 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT03985943/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT03985943/SAP_001.pdf